CLINICAL TRIAL: NCT02385266
Title: Brain Imaging-based Strategies for Treating Urological Chronic Pelvic Pain Syndrome (UCPPS) Pain
Brief Title: Treating Urological Chronic Pelvic Pain Syndrome (UCPPS) Pain
Acronym: UCPPS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was closed due to recruitment limitations
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Apkar Apkarian, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00085782; R01DK100924-01 (NIH)
Record Dates: First submitted 2015-02-26; First posted 2015-03-11 (Estimated); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Chronic Prostatitis With Chronic Pelvic Pain Syndrome
Keywords: Interstitial cystitis with Painful Bladder Syndrome; Urological Chronic Pelvic Pain Syndrome
MeSH Terms: conditions — Prostatitis | interventions — Cycloserine; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- D-Cycloserine and Acetominophen (Experimental): D-cycloserine 200mg/bid and Acetaminophen prn
  Interventions: Drug: D-Cycloserine
- Placebo and Acetominophen (Placebo Comparator): Placebo capsules (lactose)/bid and Acetaminophen prn
  Interventions: Drug: Placebo (for D-cycloserine)

INTERVENTIONS:
Drug: D-Cycloserine — Pharmaceutical intervention aimed at altering central nervous system function takes place over 4.5 months with daily use of d-Cycloserine.
  Other Names: Seromycin
  Arms: D-Cycloserine and Acetominophen
Drug: Placebo (for D-cycloserine) — Lactose filled capsules to mimic DCS 200mg capsules
  Other Names: Tylenol
  Arms: Placebo and Acetominophen

SUMMARY:
The purpose of this study is to evaluate the efficacy of D-Cycloserine versus placebo treatment in reducing pain from urological chronic pelvic pain syndrome (UCPPS).

DETAILED DESCRIPTION:
This is a double blinded, randomized control trial (RCT) over a 21 week period that aims to evaluate the treatment efficacy of placebo and D-cycloserine(DCS) in men suffering from UCPPS. The brain functional and anatomical properties associated with treatment response will also be examined.

This study will emphasize on comparing, both clinically and by brain imaging, the analgesic response to placebo in both placebo responders and non-responders in addition to a novel treatment (DCS) that targets the brain's pain mechanism for UCPPS.

Subjects will be randomized to 2 arms, in a 1:1 ratio, to a DCS medication group (n=20) and a placebo medication group (n=20). Questionnaire outcomes and brain scans will occur prior to initiating treatment and at the end of the treatment period. The actual visits required are minimized, 9 visits spread out over 21 weeks, as pain, quality of life and pill ingestion timings are collected using a secure study website accessible electronically.

ELIGIBILITY:
Inclusion Criteria:

* Males greater than 18 years of age, with no racial/ethnic restrictions;
* Meets diagnostic criteria for Interstitial Cystitis with Painful Bladder Syndrome (IC/PBS) and/or Chronic Prostatitis with Chronic Pelvic Pain Syndrome (CP/CPPS);
* Reports symptoms of discomfort or pain in the pelvic or abdominal region for at least a 3 mo period within the last 6 mo;
* Must have a Visual Analog Scale (VAS) pain score >40 mm (of 100 mm maximum) at the baseline visit (UCPPS pain moderate to severe);
* Must be in generally stable health;
* Must be willing to abstain from drinking alcohol during the course of the study;
* Must be able to read and speak English and be willing to read and understand instructions as well as questionnaires;
* Must sign an informed consent document after a complete explanation of the study documenting that they understand the purpose of the study, procedures to be undertaken, possible benefits, potential risks, and are willing to participate.

Exclusion Criteria:

* Urological pain associated with any systemic signs or symptoms, e.g., fever, chills;
* Evidence of a facultative Gram negative or enterococcus with a value of ≥ 100,000 CFU/ml in mid-stream urine (VB2);
* Has a second chronic pain condition (e.g., chronic low back pain, temporomandibular joint syndrome, etc.) that would prevent a clear interpretation of the study results;
* History of tuberculous cystitis, bladder cancer, carcinoma in situ, prostate cancer, or urethral cancer;
* History of significant pelvic comorbidities, including inflammatory bowel disease (such as Crohn's disease or ulcerative colitis), has undergone pelvic radiation, systemic chemotherapy, or intravesical chemotherapy, or has been treated with intravesical Bacillus Calmette-Guerin (BCG) or unilateral orchialgia without other pelvic symptoms, has an active urethral stricture, ureteral calculi, urethral diverticulum, or has a neurological disease or disorder affecting the bladder;
* Significant other medical conditions/diseases, such as significant renal disease or a history of renal insufficiency, unstable diabetes mellitus, congestive heart failure, coronary or peripheral vascular disease, chronic obstructive lung disease, or malignancy;
* Neurologic disorder, including history of seizures;
* Major psychiatric disorder during the past 6 months;
* Moderate or severe depression, as determined by the Hospital Anxiety and Depression Scale, or any active suicidal ideation;
* History of, or current, substance abuse/dependence including alcohol;
* Known sensitivity to D-cycloserine;
* Currently taking any of the following medications: ethionamide, dilantin, isoniazid (INH), pyridoxine (vitamin B6)
* Use of therapeutic doses of antidepressant medications (i.e., tricyclic depressants, Selective Serotonin Reuptake Inhibitor (SSRIs), Serotonin-Norepinephrine Reuptake Inhibitor (SNRIs); low doses used for sleep may be allowed), as these medications can alter pain transmission;
* Current use of low dose aspirin;
* Indication that the subject is unlikely to be compliant due to unmanaged medical or psychological condition(s), including neurological, psychological, or speech/language problems that will interfere or prevent with his understanding of consent, his ability to comply with the protocol or ability to complete the study;
* Any change in medication for urological pain in the last 30 days;
* High dose opioid prophylaxis, as defined as > 50mg morphine equivalent/day;
* Any medical condition that in the investigator's judgment may prevent the individual from completing the study or put the individual at undue risk;
* In the judgment of the investigator, unable or unwilling to follow protocol and instructions;
* Evidence of poor treatment compliance, in the judgment of the investigator;
* Intra-axial implants (e.g. spinal cord stimulators or pumps); and
* All exclusion criteria for Magnetic Resonance (MR) safety: any metallic implants, brain or skull abnormalities, tattoos on large body parts, and claustrophobia.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vania Apkarian, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Following publication of primary analyses, de-identified scan and clinical data will be posted to NIH-sponsored Open Pain database.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | D-Cycloserine and Acetominophen | Placebo and Acetominophen
Started | 12 | 12
Completed | 11 | 9
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-Cycloserine and Acetominophen | Placebo and Acetominophen | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (14.8) | 39.7 (10.3) | 43.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS)
Description: The visual analog scale (VAS) is a measurement tool used to assess the level of pain experienced by a patient. The scale is a 100 mm horizontal line, with one end representing "no pain" and the other end representing "worst pain imaginable." The patient is asked to mark on the line the point that best represents their level of pain.
  The minimum score is 0 mm, indicating no pain, while the maximum score is 100 mm, indicating the worst pain imaginable. Higher scores on the VAS indicate a worse outcome, while lower scores indicate a better outcome.
  The VAS score can be determined by measuring the distance in millimeters from the left end of the line to the point marked by the patient. The range of scores can be used to interpret the level of pain experienced by the patient, with higher scores indicating greater pain severity.
Time Frame: 18 weeks after baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-Cycloserine and Acetominophen | Placebo and Acetominophen
Number analyzed (Participants) | 11 | 9
units on a scale | 3.2 (2.6) | 3.0 (1.5)

ADVERSE EVENTS:
Arm/Group | D-Cycloserine and Acetominophen | Placebo and Acetominophen
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
The study was closed due to recruitment limitations. Given the challenges in recruitment, the investigators decided to terminate the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes